CLINICAL TRIAL: NCT06649617
Title: The Effect of Virtual Reality and Music Therapy on Physiological Parameters and Anxiety in Nursing Interventions Applied to Intensive Care Patients: A Randomized Controlled Experimental Study
Brief Title: The Effect of Virtual Reality and Music Therapy on Physiological Parameters and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Hamiyet KIZIL, PhD RN Assistant Professor Hamiyet KIZIL, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 223
Record Dates: First submitted 2024-10-09; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Pain; Anxiety; Physiological Parameter
Keywords: pain; anxiety; physiological parameter; intensive care; nursing interventions,; music threapy; virtual reality
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Standard Procedure) (Experimental): Before the application of nursing interventions ( Intramuscular , Intravenous , Subcutaneous Injection) to the patients, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State- Trait Anxiety Scale were evaluated. Then , information was given about the nursing intervention to be performed as a standard procedure . The nursing intervention was applied. After the application, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State- Trait Anxiety Scale were evaluated. Whichever nursing intervention was necessary for the patients ( Intramuscular , Intravenous , Subcutaneous Injection), that application was applied. No unnecessary procedure was applied.
  Interventions: Other: Control Group (Standard Procedure)
- Music Therapy Group (Experimental): Before the application of nursing interventions ( intramuscular , intravenous , subcutaneous injection) to the patients, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State -Trait Anxiety Scale were evaluated. During the nursing intervention, the patients were made to listen to Büzürk makam, a Turkish musical makam. After the application, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State -Trait Anxiety Scale were evaluated. Whichever nursing intervention was necessary ( intramuscular , intravenous , subcutaneous injection), that application was performed on the patients . No unnecessary procedure was performed.
  Interventions: Other: Music Therapy Group
- Virtual Reality Group (Experimental): Before the application of nursing interventions ( Intamuscular , Intravenous , Subcutaneous Injection) to the patients, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State -Trait Anxiety Scale were evaluated. During the nursing intervention, the patients watched 3D videos with relaxation effect with virtual glasses. After the application, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State -Trait Anxiety Scale were evaluated. Whichever nursing intervention was necessary ( Intamuscular , Intravenous , Subcutaneous Injection), that application was performed on the patients . No unnecessary procedure was performed.
  Interventions: Other: Virtual Reality Group

INTERVENTIONS:
Other: Control Group (Standard Procedure) — Before the application of nursing interventions ( Intramuscular , Intravenous , Subcutaneous Injection) to the patients, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State- Trait Anxiety Scale were evaluated. Then , information was given about the nursing intervention to be performed as a standard procedure . The nursing intervention was applied. After the application, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State- Trait Anxiety Scale were evaluated. Whichever nursing intervention was necessary for the patients ( Intramuscular , Intravenous , Subcutaneous Injection), that application was applied. No unnecessary procedure was applied. .
  Arms: Control Group (Standard Procedure)
Other: Music Therapy Group — Before the application of nursing interventions ( intramuscular , intravenous , subcutaneous injection) to the patients, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State -Trait Anxiety Scale were evaluated. During the nursing intervention, the patients were made to listen to Büzürk makam, a Turkish musical makam. After the application, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State -Trait Anxiety Scale were evaluated. Whichever nursing intervention was necessary ( intramuscular , intravenous , subcutaneous injection), that application was performed on the patients . No unnecessary procedure was performed.
  Arms: Music Therapy Group
Other: Virtual Reality Group — Before the application of nursing interventions ( Intamuscular , Intravenous , Subcutaneous Injection) to the patients, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State -Trait Anxiety Scale were evaluated. During the nursing intervention, the patients watched 3D videos with relaxation effect with virtual glasses. After the application, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State -Trait Anxiety Scale were evaluated. Whichever nursing intervention was necessary ( Intamuscular , Intravenous , Subcutaneous Injection), that application was performed on the patients . No unnecessary procedure was performed.
  Arms: Virtual Reality Group

SUMMARY:
Background and Aim: Invasive procedures such as intravenous , intramuscular and subcutaneous Injection practices are among the most frequently performed nursing interventions in ıntensive care units. However, although nursing interventions positively affect the clinical results of the patient, they can cause anxiety and pain. In recent years, music therapy and virtual reality, which are nonpharmacological methods, have been widely used in reducing pain and anxiety. Based on this information, this study was conducted as a randomized controlled experimental to evaluate the effects of virtual reality and music therapy on physiological parameters and anxiety in nursing ınterventions applied to ıntensive care patients.

Methods:The research was conducted with 90 patient in intensive care unit. The patients in the sample group were randomly determined by the researcher as Control Group (Standard Procedure), Music Therapy Group and Virtual Reality Group. The selection of patients included in the study was made using a random number table. Research data were collected using a structured patient information form, VAS pain scale , and state and trait anxiety inventory.The data were analyzed using SPSS 25 program.

Keywords: music therapy, virtual reality, nursing interventions, intensive care

DETAILED DESCRIPTION:
This study was conducted as a Randomized Controlled Experimental to evaluate the Effects of Virtual Reality and Music Therapy on Physiological Parameters and Anxiety in Nursing Interventions Applied to Intensive Care Patients.

Hypotheses of the Research; H1 1 : Virtual Reality and Music Therapy Improve Physiological Parameters in Nursing Interventions Applied to Intensive Care Patients.

H1 2 : Virtual Reality and Music Therapy in Nursing Interventions Applied to Intensive Care Patients reduces pain.

H1 3 : Virtual Reality and Music Therapy reduce anxiety in Nursing Interventions Applied to Intensive Care Patients .

Variables of the Research; The independent variables of the study are music therapy , virtual reality technology and standard procedure (explanation of the nursing intervention to the patient before the procedure).

The dependent variables of the study are the physiological parameters (pulse, blood pressure, fever, pain) and anxiety levels of the patients during nursing interventions.

The intensive care unit of a foundation university hospital between May 2022 and July 2022. In order to determine the number of patients constituting the research sample, a similar study (13) was taken as an example in the relevant literature and the power analysis G* Power 3.1 software was used. In this study, the sample size was calculated as 84, with 28 participants in each group, to reach a power level of 95% at a 0.5 effect size and 5% error level. Considering the high power of the test and the losses in the study , a total of 90 people were reached, 30 in each group. The patients in the sample group were randomly determined by the researcher as Control Group (Standard Procedure), Music Therapy Group and Virtual Reality Group. The selection of patients included in the study was made using a random number table. The randomization table was created by using the website http://stattrek.com/statistics/random-number-generator.aspx for randomization . As a result, the sample of the study consisted of 90 patients in total, 30 participants in each patient group, who were informed after the purpose of the study was explained and permission was obtained to participate in the study and who met the sample criteria of the study. The sample criteria were; the patient was over 18 years of age, had no visual or hearing impairment, had stable hemodynamic and physiological parameters (pulse, respiration, blood pressure, oxygen saturation , pain), was not intubated and volunteered for the study.Research data were collected using a structured patient information form, VAS pain scale , and state and trait anxiety inventory.application, the 3 groups of the study (control, virtual reality, music therapy ) were randomly assigned to 3 halls of the intensive care unit . Thus, the application was performed on one group of patients in one hall. All patients participating in the study filled out the "Structured Patient Information Form". Then, the patients were divided into 3 groups. The standard procedure (verbal procedure explanation) was applied to the control group patients. The virtual reality group patients were shown 3-dimensional videos with a relaxation effect using virtual glasses. The music therapy group patients were made to listen to the Büzürk makam , a Turkish musical makam . In this study, while nursing interventions ( Intamuscular , Intravenous , Subcutaneous Injection) were applied to all 3 groups of patients, the physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain and anxiety levels of the patients were evaluated before and after the procedure .

Application in Control Group: Before the application of nursing interventions ( Intramuscular , Intravenous , Subcutaneous Injection) to the patients, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State- Trait Anxiety Scale were evaluated. Then , information was given about the nursing intervention to be performed as a standard procedure . The nursing intervention was applied. After the application, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State- Trait Anxiety Scale were evaluated. Whichever nursing intervention was necessary for the patients ( Intramuscular , Intravenous , Subcutaneous Injection), that application was applied. No unnecessary procedure was applied. After all the applications were completed, virtual glasses or music therapy was applied to the volunteers from the control group in order to ensure the principle of equality, which is one of the ethical principles .

Application in Music Therapy Group: Before the application of nursing interventions ( intramuscular , intravenous , subcutaneous injection) to the patients, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State -Trait Anxiety Scale were evaluated. During the nursing intervention, the patients were made to listen to Büzürk makam, a Turkish musical makam. After the application, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State -Trait Anxiety Scale were evaluated. Whichever nursing intervention was necessary ( intramuscular , intravenous , subcutaneous injection), that application was performed on the patients . No unnecessary procedure was performed.

Application in Virtual Reality Group: Before the application of nursing interventions ( Intamuscular , Intravenous , Subcutaneous Injection) to the patients, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State -Trait Anxiety Scale were evaluated. During the nursing intervention, the patients watched 3D videos with relaxation effect with virtual glasses. After the application, the patients' physiological parameters (fever, pulse, blood pressure, respiration and oxygen saturation ), pain levels with VAS and anxiety levels with State -Trait Anxiety Scale were evaluated. Whichever nursing intervention was necessary ( Intamuscular , Intravenous , Subcutaneous Injection), that application was performed on the patients . No unnecessary procedure was performed.

Ethical considerations Before starting the research, permission was obtained from the Istanbul Beykent University Social and Human Sciences Scientific Research and Publication Ethics Board with the decision number 223 dated 09.05.2022. Written permission was obtained from the institution where the research was conducted. After the information about the research, the patients who agreed to participate voluntarily were asked to read and sign the consent forms prepared for each group. The researcher, who completed the application phase of the research, is a faculty member in the Department of Nursing Fundamentals.

Data analysis The data obtained in the study were obtained using SPSS (Statistical Package for Social Sciences ) for Windows 25.0 program was used for analysis. Descriptive statistical methods were used for data evaluation as number, percentage, mean, standard deviation. Differences between proportions of categorical variables in independent groups were analyzed using Chi-Square and Fisher It was analyzed with exact tests. T-test was used to compare quantitative continuous data between two independent groups. Dependent groups t-test was used to compare within-group measurements.

ELIGIBILITY:
Inclusion Criteria:

Patients;

* must be over 18 years old,
* have no visual or hearing impairment,
* have stable hemodynamic and physiological parameters (pulse, respiration, blood pressure, oxygen saturation, pain),
* be not intubated,
* be willing to participate in the study.

Exclusion Criteria:

Patients;

* have visual and hearing impairment,
* have unstable hemodynamic and physiological parameters (pulse, respiration, blood pressure, oxygen saturation, pain),
* are intubated,
* do not volunteer for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Pain severity | 2 month
  Patients were informed about the Visual Analogue Scale. Visual Analogue Scale: The level of pain, which is one of the physiological parameters, will be evaluated with the VAS pain scale . The scale includes facial expressions that show the level of pain between 0 and 10.
physiological parameter values (pulse rate /minute, respiratory rate/minute, systolic and diastolic blood pressure mm/Hg, oxygen saturation %, body temperature oC) | 2 month
  patients were informed about physiological parameters. Physiological parameter values (ulse rate /minute, respiratory rate/minute, systolic and diastolic blood pressure mm/Hg, oxygen saturation %, body temperature oC)

SECONDARY OUTCOMES:
Anxiety level | 2 month
  Patients were informed about the State-Trait Anxiety Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Hamiyet Kızıl, Phd RN, Principal Investigator — Istanbul Beykent University
Locations (1):
- Beykent University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamdan KM, Shaheen AM, Abdalrahim MS. Barriers and enablers of intensive care unit nurses' assessment and management of patients' pain. Nurs Crit Care. 2022 Jul;27(4):567-575. doi: 10.1111/nicc.12624. Epub 2021 Apr 1. PMID 33797160
- [Result] Golino AJ, Leone R, Gollenberg A, Gillam A, Toone K, Samahon Y, Davis TM, Stanger D, Friesen MA, Meadows A. Receptive Music Therapy for Patients Receiving Mechanical Ventilation in the Intensive Care Unit. Am J Crit Care. 2023 Mar 1;32(2):109-115. doi: 10.4037/ajcc2023499. PMID 36854910
- [Result] Koticha P, Katge F, Shetty S, Patil DP. Effectiveness of Virtual Reality Eyeglasses as a Distraction Aid to Reduce Anxiety among 6-10-year-old Children Undergoing Dental Extraction Procedure. Int J Clin Pediatr Dent. 2019 Jul-Aug;12(4):297-302. doi: 10.5005/jp-journals-10005-1640. PMID 31866714